CLINICAL TRIAL: NCT01421355
Title: A Pilot Study of Moderate Hyperbilirubinemia in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Mark Alan Creager, MD, Mark A. Creager, MD, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1R03DK094510-01 (NIH)
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atazanavir 300 mg BID (Experimental): Atazanavir 300 mg BID for 4 days.
  Interventions: Drug: Atazanavir

INTERVENTIONS:
Drug: Atazanavir — The study design is a single arm, open label trial. Treatment is atazanavir 300 mg BID per day for 4 days. The Brigham and Women's Hospital Investigational Drug Service (IDS) will dispense study drug.

SUMMARY:
Specific Aim: To establish the feasibility of studying the change in endothelial function caused by induced moderate hyperbilirubinemia in type 1 diabetes. Atazanavir, a drug that inhibits bilirubin conjugation, will be used to induce moderate hyperbilirubinemia. Endothelial function will be measured before and after atazanavir therapy. In addition, plasma markers of antioxidant capacity and oxidant stress will be measured as proof-of-concept that induced moderate hyperbilirubinemia has favorable effects on oxidative stress in type 1 diabetes.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is associated with a markedly increased risk of both macro- and microvascular disease. Excess pro-oxidants and insufficient antioxidants each contributes to oxidant stress in DM. Oxidant stress induces endothelial dysfunction, a major determinant of vascular damage. In DM, hyperglycemia and elevated free fatty acids (FFAs) induce generation of reactive oxygen species (ROS) by stimulating protein kinase C (PKC) and nicotinamide adenine dinucleotide phosphate (NADPH) oxidase (Figure 1). In addition, hyperglycemia activates the renin-angiotensin system, and angiotensin II (Ang II) additively stimulates PKC and NADPH oxidase.

Bilirubin, long regarded as metabolic waste, is, in fact, a potent antioxidant scavenger of ROS. It also directly inhibits both protein kinase C and the NADPH oxidase system, augmenting its antioxidant activity (Figure 1). Moreover, bilirubin inhibits Ang II-mediated vasoconstriction and ROS generation. Experimental models suggest that hyperbilirubinemia may preserve diabetes-associated endothelial function and prevent vasculopathy. Furthermore, epidemiological studies demonstrate that higher bilirubin levels are associated with a reduced risk of vascular disease in DM. Bilirubin therefore emerges as a potentially critical molecule to protect against diabetic vascular and renal damage. However, limited translational research has addressed raising bilirubin levels as a preventive therapy for vascular disease in DM.

Accordingly, the investigators seek to establish the feasibility of studying the change in endothelial function caused by induced moderate hyperbilirubinemia in type 1 diabetes. the investigators will take advantage of the recently described use of atazanavir to safely achieve moderate hyperbilirubinemia. Atazanavir is a protease inhibitor used to treat HIV infection that competitively inhibits hepatic 1A1 isoform of uridine diphosphoglucose glucuronosyltransferase (UGT1A1), limiting bilirubin clearance and inducing hyperbilirubinemia (Figure 2). This mimics Gilbert's syndrome, a benign unconjugated hyperbilirubinemia due to partial genetic deficiency of UGT1A1.

This work has the potential to identify iatrogenic moderate hyperbilirubinemia as a strategy to interrupt key mechanisms of type 1 diabetes-associated macro- and microvascular disease.

This is a physiologic study. The design is a single arm and open label. There are three study visits: a screening visit, a baseline visit, and a final visit. The treatment is atazanavir 300 mg PO bid. The treatment period is 4 days. The primary study outcome is forearm vascular function. The principal secondary outcomes are serum antioxidant defense capacity and measures of oxidant stress.

The investigators aim to study 20 subjects to completion over the 12 month funding period. The investigators anticipate enrolling 40 subjects before 20 complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of diabetes plus casual plasma glucose concentration ≥ 200 mg/dl (11.1 mmol/l), or;
2. FPG ≥ 126 mg/dl (7.0 mmol/l), or;
3. 2-h postload glucose ≥ 200 mg/dl (11.1 mmol/l) during an OGTT. In addition, subjects would be required to be at increased risk of cardiovascular events, defined as:

   * microalbuminuria, or;
   * T1DM duration of > 20 years.

Exclusion Criteria:

1. HIV infection
2. Gilbert's syndrome
3. Hepatic failure or active hepatitis,
4. Unstable cardiovascular disease, including angina, heart failure or arrhythmia
5. drug abuse including alcoholism or addiction to cocaine, heroin or amphetamines
6. Use of medications that significantly with atazanavir
7. Pregnancy, or inability to practice adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Beckman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atazanavir 300 mg BID
Started | 21
Completed | 15
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Atazanavir 300 mg BID
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Brachial Artery Diameter
Description: The primary endpoint is the difference in the change in brachial artery diameter in response to a flow stimulus at visit 2 and 3. It is anticipated that a response will occur following atazanavir therapy compared with baseline. The principal secondary endpoints are the serum measures of oxidant stress and antioxidant capacity.
Time Frame: Day 0 and Day 4
Measure: Mean (Standard Deviation); unit: percentage of dilation
Arm/Group | Atazanavir 300 mg BID
Number analyzed (Participants) | 15
percentage of dilation | -0.93 (2.4)

ADVERSE EVENTS:
Arm/Group | Atazanavir 300 mg BID
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No